CLINICAL TRIAL: NCT04167228
Title: Impact of Ceftazidime / Avibactam Treatment vs Better Available Therapy on Mortality of Patients With Infections Caused by Carbapenem-resistant Enterobacteria
Acronym: CAVICOR
Status: Completed | Type: Observational
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Other Study IDs: FCO-CAV-2018-01
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Carbapenem-Resistant Enterobacteriaceae Infection
Keywords: ceftazidime / avibactam; carbapenem resistant enterobacteria
MeSH Terms: interventions — avibactam, ceftazidime drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CRE infected patients treated with ceftazidime-avibactam: Patients with infections caused by carbapenem resistant enterobacteria treated with ceftazidime-avibactam
  Interventions: Drug: Ceftazidime-Avibactam
- CRE infected patients treated with best available treatment: Patients with infections caused by carbapenem resistant enterobacteria treated with the best available treatment
  Interventions: Drug: Best Available Therapy

INTERVENTIONS:
Drug: Ceftazidime-Avibactam — Patients with complicated urinary tract infections, nosocomial pneumonia (including pneumonia associated with ventilation), complicated intra-abdominal infections or bacteremia (if the focus of infection is any of the above, the patient should be included in both groups) due to CRE, treated > 2 days with ceftazidime-avibactam.
  Groups: CRE infected patients treated with ceftazidime-avibactam
Drug: Best Available Therapy — Patients with complicated urinary tract infections, nosocomial pneumonia (including pneumonia associated with ventilation), complicated intra-abdominal infections or bacteremia (if the focus of infection is any of the above, the patient should be included in both groups) due to CRE, treated > 2 days with the best available treatment other than ceftazidime-avibactam.
  Groups: CRE infected patients treated with best available treatment

SUMMARY:
Patients with infections caused by carbapenem-resistant enterobacteria treated with CAZ-AVI versus patients treated with BAT are compared. The BAT group includes fosfomycin, tigecycline, gentamicin, meropenem and colistin.

DETAILED DESCRIPTION:
Carbapenem-resistant enterobacteria (CRE) are a public health problem. The morbidity and mortality of patients with invasive infections due to CRE are high. The best treatment is unknown, however, combination therapy with at least 2 active drugs is often recommended for high-risk patients, and monotherapy is probably not inferior to this in low-risk patients.

Ceftazidime-avibactam is active against many CRE, and in some countries it has been prescribed under compassionate use programs for these infections; It has recently been approved by the FDA and the EMA for specific indications. Recent data suggest that ceftazidime-avibactam may be superior for the treatment of infections caused by sensitive CRE, rather than traditional regimens that often include colistin, usually combined with other drugs. However, these studies include a low number of patients and are subject to important biases.

Additionally, the development of resistance to this drug during / after treatment has been described and is worrying.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complicated urinary tract infections, nosocomial pneumonia (including pneumonia associated with ventilation), complicated intra-abdominal infections or bacteremia (if the focus of infection is any of the above, the patient should be included in both groups) due to CRE, treated > 2 days with ceftazidime-avibactam. Patients with bacteremia can be included in one of the other cohorts if the focus of the infection is the urinary tract, respiratory tract or an intra-abdominal infection and they meet the appropriate criteria (see below). The retrospective design of this study has been carried out to avoid the induction of the prescription of ceftazidime-avibactam in each center. For this, patients will be included at the end of the period of evaluation of the primary objective (crude mortality at day 30). If more than one patient can be used as a control, the one with the closest admission date will be chosen.

Control: local historical cohort - Patients treated with ceftazidime-avibactam will be compared with patients treated with BAT. Because after approval of the use of ceftazidime-avibactam, BAT could be used less frequently to treat this type of infection, patients treated with BAT from January 1, 2014 will be included. These patients will be matched by hospital, type of hospital. infection (urinary tract vs others) and INCREMENT score.

Exclusion Criteria:

* The infection is considered polymicrobial according to the standard microbiological interpretation of the crop results (except for complicated intra-abdominal infections, in which case, polymicrobial infections are allowed).
* Patients with infections caused by CRE without susceptibility to ceftazidime-avibactam.
* The patient is participating in a clinical trial that involves active treatment for infections.
* Patients with cardiopulmonary no resuscitation order or with a life expectancy < 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with infections caused by carbapenem resistant enterobacteria
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
30-day mortality rate | At day 30 after the start of the treatment
  To describe the 30-day mortality rate in the caz-avi group and in the group with the best available therapy of patients with infections caused by carbapenem-resistant enterobacteria.
Clinical response on day 21 | At day 21 after the start of the treatment
  To describe the clinical response on day 21 of the caz-avi group and in the group with the best available therapy of patients with infections caused by carbapenem-resistant enterobacteria.

SECONDARY OUTCOMES:
Microbiological response | At day 30 after the start of the treatment
  Microbiological response in the Test-of-cure, categorized as eradication, microbiological failure or uncertain.
30-day mortality rate in the group of patients with caz-avi in monotherapy and in the group with combined therapy with caz-avi | At day 30 after the start of the treatment
  Describe the 30-day mortality rate in the group of patients with caz-avi in monotherapy and in the group with combined therapy with caz-avi, who present with infections caused by carbapenem-resistant enterobacteria.
Risk factors associated with the development of resistance to ceftazidime-avibactam during treatmen | At day 30 after the start of the treatment
  Describe the rates and risk factors associated with the development of resistance to ceftazidime-avibactam (MIC> 8 microg / mL) during treatment
Duration of hospital stay after infection | At day 30 after the start of the treatment
  Number of days elapsed from the end of antibiotic treatment until discharge and duration of ICU stay if appropriate.
Duration of antibiotic treatment during the episode | At day 30 after the start of the treatment
  Number of days of antibiotic treatment during the episode
Recurrence | At day 30 after the start of the treatment
  Reappearance of the infection according to the same criteria and by the same microorganism
Safety evaluation of the treatment | At day 30 after the start of the treatment
  Number of adverse reactions related to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Juan José Castón Osorio, MD, Principal Investigator — Hospital Universitario Reina Sofía
Locations (17):
- Spain (17):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Gran Canaria "Dr. Negrín", Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Complejo Hospitalario Universitario A Coruña, A Coruña, Coruña
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Clínico de Barcelona, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
The information collected will be of public access by request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the trial results are public.
Access Criteria: By request to uicec@imibic.org